CLINICAL TRIAL: NCT06528444
Title: Randomized, Double-blind, Multicenter, Phase III Clinical Trial Evaluating the Efficacy and Safety of Dexamethasone Compared to Placebo in Patients With Severe Influenza
Brief Title: Clinical Trial Evaluating the Efficacy and Safety of Dexamethasone Compared to Placebo in Patients With Severe Influenza
Acronym: FLUDEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria y Biomédica de Alicante (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FLUDEX
Record Dates: First submitted 2024-07-11; First posted 2024-07-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): placebo 1 capsule (6 mg) /day for 7 days.
  Interventions: Drug: Grup 1 placebo
- dexamethasone (Active Comparator): dexamethasone 1 capsule (6 mg)/day for 7 days
  Interventions: Drug: Grup 2 dexametasona

INTERVENTIONS:
Drug: Grup 1 placebo — placebo 1 capsule (6 mg) /day for 7 days.
  Arms: Placebo
Drug: Grup 2 dexametasona — dexamethasone 1 capsule (6 mg)/day for 7 days
  Arms: dexamethasone

SUMMARY:
Clinical trial with an active ingredient of a pharmaceutical specialty marketed in Spain vs. placebo.

Randomized, double-blind, multicenter phase III clinical trial that evaluates the efficacy and safety of dexamethasone compared to placebo in patients with severe influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years.
2. Diagnosis of influenza A or B virus infection by antigen or RT-PCR (local laboratory) at the time of entry or at 48 hours prior to randomization in respiratory specimens (nasopharyngeal swab or bronchoalveolar lavage).
3. Hospitalized patients with an estimated hospital stay of more than 24 hours.
4. In previous treatment or concomitant start of treatment with oseltamivir.
5. For women of childbearing age, use of contraceptive methods until day 30 after completion of treatment.
6. Signed informed consent.

Exclusion Criteria:

* 1. Patients with bronchial hyperresponsiveness that requires systemic corticosteroids for more than 24 hours.

  2. Pre-inclusion treatment with corticosteroids for more than 24 hours at a dose equal to or higher than 1 mg/kg methyl-prednisolone (0.2 mg/kg dexamethasone or 1.25 mg/kg prednisone).

  3. Inability to administer oral oseltamivir. 4. Patients on ECMO (extracorporeal membrane oxygenation). 5. Pre-existing condition or use of medication that, in the opinion of the local investigator, may pose a risk for the administration of corticosteroids.

  6. Patients with severe comorbidity with life expectancy of less than six months in the opinion of the investigator.

  7. Patients co-infected with SARS-CoV-2 or RSV.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
To compare the percentage of patients hospitalized | 10 days
  To compare the percentage of patients hospitalized with influenza according to treatment arm (oseltamivir-dexamethasone vs oseltamivir-placebo) with status 3 or higher according to the Hospital Recovery Scale (status 3: hospitalization with supplemental oxygen, or 4: ICU admission without invasive mechanical ventilation, or 5: with invasive mechanical ventilation, or 6: death) on day 7 after the start of treatment.

SECONDARY OUTCOMES:
The National Early Warning Score | 10 days
  To compare the time, in days, between initiation of treatment and clinical stability according to the NEWS2<2 scale for 24 hours or until hospital discharge, taking the value of the first of the two events to occur
Common Terminology Criteria for Adverse Events (CTCAE) scale | 10 days
  To compare the frequency of serious adverse effects between groups (grades 3, 4 and 5 on the CTCAE scale).
Rate of metabolic impact of dexamethasone | 10 days
  To evaluate the metabolic impact of dexamethasone by comparing the function of occurrence of sustained hyperglycemia level 1 and 2, and episodes of hyperglycemia during and at the end of dexamethasone treatment.
the average hospital stay | 10 days
  To compare the average hospital stay (expressed in days) according to treatment group.
Number of pacients in ICU admission | 10 days
  To compare the function of occurrence over time of clinical failure, defined as progression to: need for ICU admission, need for intubation or death.
mortality | 90 days
  To compare mortality at days 10, 30 and 90 post-randomization.
the impact of treatment Barthel Index | 90 days
  To evaluate the impact of treatment on dependency (Barthel Index) at the time of discharge or at the end of treatment, and at 30 and 90 days after randomization.
  The final score ranges from 0 to 100, with 100 being the maximum independence and 0 being the maximum dependence.
the impact of treatment Clinical Frailty Score | 90 days
  To evaluate the impact of treatment on frailty (Clinical Frailty Score) at the time of discharge or at the end of treatment, and at 30 and 90 days after randomization.
  . level descriptions and their corresponding labels. Most notably, CFS level 2 changed from "Well" to "Fit", level 4 from "Vulnerable" to "Living with Very Mild Frailty", and levels 5-8 were restated as "Living with..." mild, moderate, severe, and very severe frailty, respectively
To evaluate the impact of steroid treatment on the evolution of the nasal microbiome expressed in alpha diversity. | 10 days
  To evaluate the impact of steroid treatment on the evolution of the nasal microbiome expressed in alpha diversity.
  Using NGS and then the consecutive bioinformatic analysis. More specifically, the alpha diversity would be the result of the Shannon Index and the number of ASVs (Amplicon sequence variant).
the kinetics of influenza virus in nasopharyngeal swabs using Ct | 10 days
  To evaluate the kinetics of influenza virus in nasopharyngeal swabs (using Ct and ) in both groups.
the kinetics of influenza virus in nasopharyngeal swabs using viral quantification per human cell | 10 days
  To evaluate the kinetics of influenza virus in nasopharyngeal swabs (viral quantification per human cell) in both groups.
Evaluation inflammatory markers CRP | 10 days
  Evaluation the impact of treatment on inflammatory markers CRP
Evaluation inflammatory markers PCT | 10 days
  Evaluation the impact of treatment on inflammatory markers PCT
Evaluation inflammatory markers IL-6 | 10 days
  Evaluation the impact of treatment on inflammatory markers IL-6
Evaluation inflammatory markers IL-10 | 10 days
  Evaluation the impact of treatment on inflammatory markers IL-10

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital General Universitario Dr. Balmis de Alicante (centro coordinador), Alicante
  - Hospital General Universitario de Elche, Elche

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramos-RIncon JM, Cebollada J, Giner L, Paz Ventero M, Moreno-Perez O, Otero-Rodriguez S, Sanchez-Paya J, Rodriguez JC, Merino E. Efficacy and safety of dexamethasone compared to placebo in patients with severe influenza infection. (FLUDEX study): a study protocol for a randomised controlled trial in Spain. BMJ Open. 2025 Sep 26;15(9):e103119. doi: 10.1136/bmjopen-2025-103119. PMID 41005772